CLINICAL TRIAL: NCT00880984
Title: Compression Anastomosis Using the CAR™ 27
Brief Title: Compression Anastomosis Using the Compression Anastomosis Ring (CAR™ 27)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: novoGI (Industry)
Responsible Party: Prof. Spyros Papavramidis, AHEPA university Hospital of Thessaloniki
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-CAR-07-Gr-01
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Surgery
Keywords: Colon Anastomosis; Rectum Anastomosis; Intestine; Colorectal Surgery; Colorectal Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Compression Anastomosis Ring: CAR™ 27 — Creation of anastomosis in colorectal surgeries using CAR™ 27
  Other Names: CAR™ 27

SUMMARY:
Purpose:

Evaluation of the CAR™ 27 for the creation of compression anastomoses.

Indication:

Compression Anastomosis Ring (CAR™ 27) device for creation of circular anastomoses during colonic or colorectal resection.

Study Design:

Prospective, open labeled study.

Patient Population:

Male or female subjects 18 years of age or older who are scheduled for non emergency laparoscopic or open colonic or colorectal resections. A temporary loop ileostomy/colostomy can be preformed up to the discretion of the surgeon.

No. of Subjects:

15 patients estimated up to three months to enroll.

Duration of Treatment:

During the operation - creation of the anastomosis.

Duration of Follow-up:

Follow-up evaluation will be performed daily while hospitalized, during a post-op clinic visit at approximately 1 month (30 days ± 5 days) including a proctoscopic exam and by phone after 3 months.

Endpoints:

To evaluate the creation of a safe and functioning anastomosis and the occurrence of adverse events related to the use of the CAR™ 27 device.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old.
2. Patient is scheduled for a non-emergency procedure.
3. Subject signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures.

Exclusion Criteria:

1. Patient has an allergy to nickel.
2. Patient has a diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, carcinomatosis or extensively spread inflammatory bowel disease.
3. Patient is participating in another clinical trial which may affect this study's outcomes.
4. Patient has been taking regular steroid medication.
5. Patient has contraindications to general anesthesia.
6. Patient has preexisting sphincter problems or evidence of extensive local disease in the pelvis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Complications during and post procedure including leaks, bleeding, strictures, device failure, re admission, re operation, extra colonic complications etc | 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Spiros Papavramidis, Prof., Principal Investigator — AHEPA University Hospital of Thessaloniki
Locations (1):
- AHEPA University Hospital of Thessaloniki, Thessaloniki, Greece